CLINICAL TRIAL: NCT05279651
Title: Ivabradine for PREVENTion of Myocardial Injury After Noncardiac Surgery
Brief Title: Ivabradine for Prevention of Myocardial Injury After Noncardiac Surgery Trial (PREVENT-MINS)
Acronym: PREVENT-MINS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: Population Health Research Institute (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wojciech Szczeklik, Principal Investigator Wojciech Szczeklik MD PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREVENT-MINS
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Injury After Noncardiac Surgery (MINS); Myocardial Ischemia
Keywords: Myocardial ischemia; Randomized controlled trial; Blinded; Noncardiac surgery; Cardiovascular events; Myocardial injury after non-cardiac surgery; Perioperative myocardial injury; Perioperative myocardial infarction; Perioperative medicine; Heart rate; Ivabradine; Cardiovascular Diseases; Troponin; Perioperative care; Physiological Effects of Drugs; Cardiovascular Agents; Cardiac Chronotropy; Heart Rate Control
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases | interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivabradine (Active Comparator): Patients fulfilling haemodynamic requirements (i.e. systolic blood pressure ≥90 mmHg and sinus rhythm with a heart rate ≥65 beats per minute) will receive 5mg of oral ivabradine at least 1 hour before surgery and the first postoperative dose in the evening or in the morning after surgery, at least 12 hours after the preoperative dose. Starting on the day after surgery, patients will receive 5mg oral ivabradine twice a day and continue this treatment for 7 days after surgery or until hospital discharge.
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator): Patients fulfilling haemodynamic requirements (i.e. systolic blood pressure ≥90 mmHg and sinus rhythm with a heart rate ≥65 beats per minute) will receive matching placebo at least 1 hour before surgery and the first postoperative dose in the evening or in the morning after surgery, at least 12 hours after the preoperative dose. Starting on the day after surgery, patients will receive matching placebo twice a day and continue this treatment for 7 days after surgery or until hospital discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Patients fulfilling haemodynamic requirements (i.e. systolic blood pressure ≥90 mmHg and sinus rhythm with a heart rate ≥65 beats per minute) will receive 5mg of oral ivabradine at least 1 hour before surgery and the first postoperative dose in the evening or in the morning after surgery, at least 12 hours after the preoperative dose. Starting on the day after surgery, patients will receive 5mg oral ivabradine twice a day and continue this treatment for 7 days after surgery or until hospital discharge.
  Arms: Ivabradine
Drug: Placebo — Patients fulfilling haemodynamic requirements (i.e. systolic blood pressure ≥90 mmHg and sinus rhythm with a heart rate ≥65 beats per minute) will receive matching placebo at least 1 hour before surgery and the first postoperative dose in the evening or in the morning after surgery, at least 12 hours after the preoperative dose. Starting on the day after surgery, patients will receive matching placebo twice a day and continue this treatment for 7 days after surgery or until hospital discharge.
  Arms: Placebo

SUMMARY:
This study is a multicentre, randomized controlled trial of ivabradine versus placebo.

DETAILED DESCRIPTION:
The PREVENT-MINS study is a 2,500 patient multicentre, superiority randomized controlled trial of ivabradine versus placebo. The primary objective of the trial is to determine the impact of ivabradine versus placebo on the risk of MINS in patients with or at risk of atherosclerotic disease who are followed for 30 days after noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing noncardiac surgery
2. ≥45 years of age
3. Expected to require at least an overnight hospital admission after surgery
4. Provide written informed consent to participate in the PREVENT-MINS Trial, AND
5. Fulfill ≥1 of the following 5 criteria (A-E):

A. History of coronary artery disease B. History of peripheral arterial disease C. History of stroke D. Undergoing major vascular surgery, OR

E. Any 3 of 9 risk criteria:

i. Undergoing major surgery ii. History of congestive heart failure iii. History of a transient ischaemic attack iv. Diabetes and currently taking an oral hypoglycemic agent or insulin v. Age ≥70 years vi. History of hypertension vii. Serum creatinine >175 µmol/L (>2.0 mg/dl) viii. History of smoking within 2 years of surgery ix. Undergoing emergent/urgent surgery

Exclusion Criteria:

1. Conduction abnormalities:

   A. Non-sinus rhythm on ECG B. Sinoatrial or AV (2nd and 3d degree) blocks C. Sick sinus syndrome D. Long QT syndrome E. Pacemaker dependent
2. Transplanted heart (or on waiting list)
3. Use of a selected class I or III antiarrhythmic drug (quinidine, disopyramide, sotalol, ibutilide, amiodarone) or diltiazem/verapamil
4. Resting heart rate <65 beats per minute on the day of surgery
5. Systolic blood pressure <90 mmHg on the day of surgery
6. Acute decompensated heart failure, cardiogenic shock, acute myocarditis
7. Acute coronary syndrome within 2 months before surgery;
8. Stroke or transient cerebral ischaemia within 1 month before surgery
9. Known severe liver or kidney disease (MDRD creatinine clearance <15 mL/min)
10. Inability to tolerate oral intake
11. Recent use of ivabradine (<1 month)
12. Known allergy or hypersensitivity to ivabradine
13. Low-risk surgical procedure based on individual physician's judgment
14. Investigator considers the patient unreliable regarding requirement for study compliance
15. Women of childbearing potential who are not taking effective contraception, pregnant or breast-feeding
16. Previously enrolled in the PREVENT-MINS study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2146 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
MINS | 30 days after randomization
  Number of patients who experience myocardial injury after non-cardiac surgery (MINS) defined as any myocardial infarction and any elevated postoperative cardiac troponin judged as resulting from myocardial ischaemia during or within 30 days after noncardiac surgery.

SECONDARY OUTCOMES:
A composite of vascular death, non-fatal MINS, non-fatal stroke, and non-fatal cardiac arrest | 30 days after randomization
  Number of patients who have at least one of the following: vascular death, non-fatal MINS, non-fatal stroke, and non-fatal cardiac arrest
MINS not fulfilling the 4th universal definition of myocardial infarction | 30 days after randomization
  Number of patients who experience MINS not fulfilling the 4th universal definition of myocardial infarction
Myocardial infarction | 30 days after randomization
  Number of patients who experience a myocardial infarction
Vascular death | 30 days after randomization
  Number of patients who die of vascular cause
Stroke | 30 days after randomization
  Number of patients who experience a stroke
All-cause mortality | 30 days after randomization
  Number of patients who die of any cause
Days alive and at home | 30 days after randomization
  Average number of days when a patient is alive and out of hospital within 30 days after randomization
Health-related quality of life | 30 days after randomization
  Average health-related quality of life (based on EuroQol 5 Dimension, five-level version [EQ-5D])
Clinically important atrial fibrillation | 30 days after randomization
  Number of patients who experience clinically important atrial fibrillation
Clinically significant bradycardia | 30 days after randomization
  Number of patients who experience clinically significant bradycardia
Clinically significant hypotension | 30 days after randomization
  Number of patients who experience clinically significant hypotension
Phosphenes | 30 days after randomization
  Number of patients who experience phosphenes
Cancellation or postponement of surgery due to concerns about patient's heart rate | 30 days after randomization
  Number of surgeries cancelled or postponed due to heart rate concerns
Peak troponin concentration | 30 days after randomization
  Peak troponin concentration during the index hospitalization
Area under the curve troponin | 30 days after randomization
  Area under the curve of troponin concentrations measured during the hospitalization
Intraoperative mean arterial pressure | 30 days after randomization
  Intraoperative mean arterial pressure measured during the index surgery to calculate the average intraoperative mean arterial pressure
Intraoperative heart rate | 30 days after randomization
  Intraoperative heart rate measured during the index surgery to calculate the average heart rate

OTHER OUTCOMES:
Cardiac revascularization | 30 days after randomization
  Number of patients who undergo cardiac revascularization
Re-hospitalization for vascular reasons | 30 days after randomization
  Number of patients re-hospitalized for vascular reasons
Acute myocardial injury according to Fourth Universal Definition of Myocardial Infarction | 30 days after randomization
  Number of patients who experience an acute myocardial injury according to Fourth Universal Definition of Myocardial Infarction
Non-fatal cardiac arrest | 30 days after randomization
  Number of patients who experience non-fatal cardiac arrest
Acute congestive heart failure | 30 days after randomization
  Number of patients who experience acute congestive heart failure
Any symptomatic or asymptomatic episode of deep vein thrombosis or pulmonary embolism | 30 days after randomization
  Number of patients who experience any (symptomatic or asymptomatic) episode of deep vein thrombosis or pulmonary embolism
International Society on Thrombosis and Haemostasis (ISTH) major bleeding | 30 days after randomization
  Number of patients who experience major bleeding (as defined by ISTH)
BIMS | 30 days after randomization
  Number of patients who experience bleeding independently associated with mortality after noncardiac surgery (BIMS)
Infection/Sepsis | 30 days after randomization
  Number of patients who experience infection/sepsis
Acute kidney injury fulfilling Kidney Disease Improving Global Outcomes (KDIGO) criteria | 30 days after randomization
  Number of patients who experience an acute kidney injury (fulfilling KDIGO criteria)
Acute kidney injury requiring dialysis | 30 days after randomization
  Number of patients who experience an acute kidney injury requiring dialysis
Amputation | 30 days after randomization
  Number of patients who undergo an amputation
Days outside of intensive care unit | 30 days after randomization
  Average number of days alive outside of intensive care/cardiac care unit within 30 days after randomization
Length of hospital stay | 30 days after randomization
  Average length of hospital stay
Length of intensive care unit stay | 30 days after randomization
  Average length of intensive care unit stay
Discharge destination from the hospital | 30 days after randomization
  Number of patients discharge to home/long-term care facility/other
All-cause mortality | 1 year after randomization
  Number of patients who die of any cause
Vascular death | 1 year after randomization
  Number of patients who die of vascular cause
Myocardial infarction | 1 year after randomization
  Number of patients who experience a myocardial infarction
Cardiac revascularization | 1 year after randomization
  Number of patients who undergo cardiac revascularization
Non-fatal cardiac arrest | 1 year after randomization
  Number of patients who experience non-fatal cardiac arrest
Stroke | 1 year after randomization
  Number of patients who experience a stroke
Health-related quality of life | 1 year after randomization
  Average health-related quality of life (based on EuroQol 5 Dimension, five-level version [EQ-5D])
Amputation | 1 year after randomization
  Number of patients who have an amputation
Re-hospitalization for vascular reasons | 1 year after randomization
  Number of patients who experience a re-hospitalization for vascular reasons

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Szczeklik, Professor, Principal Investigator — Centre for Intensive Care and Perioperative Medicine, Jagiellonian University Medical College
Locations (26):
- Poland (26):
  - Szpital Uniwersytecki nr 1 im. dr Antoniego Jurasza w Bydgoszczy, Bydgoszcz
  - Specjalistyczny Szpital Wojewódzki w Ciechanowie, Ciechanów
  - ZZOZ Szpital Śląski w Cieszynie, Cieszyn
  - Uniwersyteckie Centrum Kliniczne Gdańskiego Uniwersytetu Medycznego, Gdansk
  - Szpital Specjalistyczny św. Łukasza w Końskich, Gmina Końskie
  - Uniwersyteckie Centrum Kliniczne im. Prof. Kornela Gibińskiego Śląski Uniwersytet Medyczny, Katowice
  - Szpital św. Rafała w Krakowie, Krakow
  - 5 Wojskowy Szpital Kliniczny z Polikliniką Samodzielny Publiczny Zakład Opieki Zdrowotnej w Krakowie, Krakow
  - Szpital Zakonu Bonifratrów św. Jana Grandego w Krakowie, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie sp. z o.o., Krakow
  - Szpital Specjalistyczny im. Stefana Żeromskiego w Krakowie, Krakow
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny 1 w Lublinie, Lublin
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 Pomorskiego Uniwersytetu Medycznego, Szczecin
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 Pomorskiego Uniwersytetu Medycznego, Szczecin
  - Specjalistyczny Szpital im. Edwarda Szczeklika w Tarnowie, Tarnów
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego Szpital Kliniczny Dzieciątka Jezus, Warsaw
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego Centralny Szpital Kliniczny, Warsaw
  - Wojskowy Instytut Medyczny Centralny Szpital Kliniczny MON, Warsaw
  - Uniwersytecki Szpital Kliniczny we Wrocławiu, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanisława Szyszko Śląskiego Uniwersytetu Medycznego w Katowicach, Zabrze
  - Szpital Uniwersytecki im. Karola Marcinkowskiego w Zielonej Górze, Zielona Góra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szczeklik W, Fronczek J, Putowski Z, Wludarczyk A, Gorka J, Seczynska B, Gryszowka D, Widawska A, Bialka S, Palaczynski P, Borys M, Kutnik P, Czarnik T, Krolicki T, Szczepanska A, Hajder N, Mozanski M, Onichimowski D, Kotfis K, Trzebicki J, Sadowski L, Solek-Pastuszka J, Grudzien P, Mudyna W, Misiewska-Kaczur A, Owczuk R, Kudlinski B, Studzinska D, Pawlik J, Makowski A, Zietkiewicz M, Przydacz M, Gozdzik W, Gola W, Jasiewicz P, Zhao Z, Shyr Y, Devereaux PJ. Ivabradine for prevention of myocardial injury after noncardiac surgery (PREVENT-MINS trial): study protocol for a randomized controlled trial. Trials. 2025 Nov 21;26(1):533. doi: 10.1186/s13063-025-09087-z. PMID 41272750
- [Derived] Szczeklik W, Fronczek J, Putowski Z, Wludarczyk A, Gorka J, Seczynska B, Gryszowka D, Widawska A, Bialka S, Palaczynski P, Borys M, Kutnik P, Czarnik T, Szczepanska A, Mozanski M, Mieszkowski M, Kotfis K, Trzebicki J, Sadowski L, Solek-Pastuszka J, Grudzien P, Mudyna W, Misiewska-Kaczur A, Owczuk R, Kudlinski B, Studzinska D, Pawlik J, Makowski A, Zietkiewicz M, Przydacz M, Gozdzik W, Gola W, Jasiewicz P, Zhao Z, Shyr Y, Devereaux PJ; PERI-CRIT Investigators. Ivabradine in Patients Undergoing Noncardiac Surgery: A Randomized Controlled Trial. Circulation. 2025 Oct 21;152(16):1126-1135. doi: 10.1161/CIRCULATIONAHA.125.076704. Epub 2025 Aug 30. PMID 40884771